CLINICAL TRIAL: NCT00846690
Title: Comparative Efficacy of 20% Benzocaine Versus TAC Alternate Gel for Control of Pain of Dental Needle Insertion in the Palate
Brief Title: Comparative Efficacy of 20% Benzocaine Versus TAC Alternate Gel
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Femme Ambrosio, University of Texas Health Science Center Houston
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-DB-08-0484
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Dental Pain; Postoperative Pain
Keywords: topical anesthetics; topical anesthesia; 20% benzocaine; TAC alternate gel; combination topical anesthetics; dental anesthesia
MeSH Terms: conditions — Toothache; Pain, Postoperative | interventions — Benzocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benzocaine (Active Comparator): serves as "active" control
  Interventions: Drug: benzocaine
- TAC (Experimental): serves as comparator
  Interventions: Drug: TAC alternate gel

INTERVENTIONS:
Drug: benzocaine — 20% benzocaine., topical placement onto site, minimal amount, for 1 minute
  Other Names: Hurricaine
  Arms: Benzocaine
Drug: TAC alternate gel — use 1 pump, place topically onto site, leave for 1-3 minutes
  Other Names: 20% TAC alternate gel
  Arms: TAC

SUMMARY:
The project is a study comparing the effectiveness of two topical anesthetics for control of pain associated with dental needle insertion in the palatal mucosa. A standard dental topical anesthetic (20% benzocaine) will serve as an "active" control and will be compared to a combination topical anesthetic, consisting of 20% lidocaine, 4% tetracaine and 2% phenylephrine (TAC Alternate Gel, Compounding Arts Pharmacy, Lafayette, LA).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers 18 years or older
2. Ability to consent to participate in the research
3. Ability to communicate a VAS score
4. Generally healthy, ASA I and ASA II
5. No known drug allergies
6. Ability to tolerate pulse oximeter and blood pressure cuff without psychological, or physiological consequence

Exclusion Criteria:

1. Allergy or other contraindications to the topical anesthetics
2. Inability to consent to participation in the study
3. Use of analgesics prior to the procedure
4. Vulnerable populations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-03 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale score | pre-op, insertion, every minute post-op for 10 minutes

SECONDARY OUTCOMES:
blood pressure | three times pre-op, insertion, ten times post-op
oxygen saturation | three times pre-op, insertion, ten times post-op
heart rate | three times pre-op, insertion, ten times post-op

CONTACTS AND LOCATIONS:
Overall Officials: Femme L Ambrosio, DDS, Principal Investigator — UT Health Science Center Houston; Arthur H Jeske, DDS, PhD, Study Chair — UT Health Science Center Houston
Locations (1):
- UT Pediatric Dentistry Clinic Houston Medical Center, 6655 Travis Suite 460, Texas, United States